CLINICAL TRIAL: NCT05861739
Title: The Effect of the Self-Care Support Program Applied to Women With Endometriosis on Quality of Life, Self-Care Behaviors, Depression, Anxiety and Stress Level
Brief Title: The Effect of the Self-Care Support Program on Women With Endometriosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 150
Record Dates: First submitted 2023-04-27; First posted 2023-05-17 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Endometriosis; Quality of Life; Depression; Anxiety; Stress
Keywords: Endometriosis; Self-care support program; Quality of Life; Motivational interview; Self-care behaviors
MeSH Terms: conditions — Endometriosis; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Endometriosis Self Care Support Program (Endometriosis Training and Motivational Interview) will be applied to the women in the intervention group.
  Interventions: Behavioral: Endometriosis Self-care Support Program
- Control group (No Intervention): Women in the control group will receive standard treatment. Training and motivational interviewing will not be applied.

INTERVENTIONS:
Behavioral: Endometriosis Self-care Support Program — ESSP will be applied to the women in the intervention group in four sessions, one week apart. In the first and second sessions, a self-care training program will be applied. In the third and fourth sessions, motivational interview will be made by contacting the women by phone.
  Arms: Intervention group

SUMMARY:
This study, was aimed to evaluate the effect of self-care support program (self-care training in endometriosis + motivational interview) applied to women with endometriosis on quality of life, self-care behaviors, depression, anxiety and stress levels.

DETAILED DESCRIPTION:
This study is a randomized controlled experimental study conducted to evaluate the effect of self-care support program applied to women with endometriosis on quality of life, self-care behaviors, depression, anxiety and stress levels.The research was carried out with the participation of two groups. Endometriosis Self-care Support program-ESSP (intervention group) will be applied to one of the groups, while the other group (control group) will receive standard treatment within the scope of the hospital protocol. Then, women's quality of life, self-care behaviors, depression, anxiety and stress levels will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive age (between 18-49 years old),
* Diagnosed with endometriosis (symptomatic patients),
* Having no medical or gynecological problems other than endometriosis,
* Literate,
* Mobile phone user,
* Non-pregnant,
* No communication barrier
* Not diagnosed with a psychiatric illness,
* Who volunteered to participate in the research,
* Women who can speak and understand Turkish will be included.

Exclusion Criteria:

* Who could not attend any session of ESSP (only in the intervention group),
* Filling the data collection forms incompletely,
* Pregnant at the time of the study and
* Women who have been hospitalized and/or had surgical operations for gynecological and medical reasons will be excluded.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Self-Care Behaviors Scale in Endometriosis | Self-care behaviors will be evaluated at the first interview, 1st and 4th months. The change in the difference between the groups in terms of self-care behaviors over time will be evaluated.
  This scale will be developed to measure the self-care behaviors of women with endometriosis.After the reliability and validity analyzes of the scale, the sub-dimensions of the scale, the number of items and the total score will be determined.
Endometriosis Health Profile | Quality of life will be evaluated at the first interview, 1st and 4th months. The variation of the difference between the groups in terms of quality of life over time will be evaluated.
  The Endometriosis Health Profile, consists of 11 questions. The lowest score that can be obtained from the entire questionnaire is 0 (best health condition), the highest score is 100 (worst health condition). The higher the score obtained from the questionnaire, the lower the quality of life.
Depression, Anxiety and Stress Scale | Depression, anxiety and stress levels will be evaluated at the first interview, 1st and 4th months. The variation of the difference between the groups in terms of depression, anxiety and stress levels over time will be evaluated.
  This scale, participants' depression, anxiety and stress levels will be evaluated.The scale consists of 21 items and 3 sub-dimensions (depression, anxiety and stress). There is a separate total score for each sub-dimension. As the score obtained from the subscale increases, the level of depression, anxiety and stress increases.

SECONDARY OUTCOMES:
Numerical Pain Scale | The pain level will be evaluated at the first interview, 1st and 4th months. The variation of the difference between the groups in terms of pain level over time will be evaluated.
  It will be used to determine the pain levels of the participants.It starts with the absence of pain (0) on numerical scales and reaches the level of unbearable pain (10).

CONTACTS AND LOCATIONS:
Overall Officials: Nurdan Demirci, Prof., Study Director — Marmara University
Locations (1):
- Marmara University, Istanbul, Başıbüyük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No